CLINICAL TRIAL: NCT02017327
Title: Safety and Efficacy Assessment of Monoprost® in Comparison With Lumigan® 0.01% and Lumigan® 0.03% Unit Dose, in Patients With Primary Open Angle Glaucoma or Ocular Hypertension, Stabilized by Lumigan® 0.01% With Ocular Surface Intolerance
Brief Title: Safety and Efficacy Assessment of Monoprost® in Comparison With Lumigan® 0.01 % and Lumigan® 0.03% Unit Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT2345-PIV-02/13; 2013-001250-10 (EudraCT Number)
Record Dates: First submitted 2013-12-02; First posted 2013-12-20 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-02

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Monoprost (Experimental): 1 drop in each eye once daily at 9.00 pm (± 1 hour) for 3 months.
  Interventions: Drug: Monoprost
- Lumigan 0.01% (Active Comparator): 1 drop in each eye once daily at 9.00 pm (± 1 hour) for 3 months.
  Interventions: Drug: Lumigan 0.01%
- Lumigan 0.03% Unit Dose (Active Comparator): 1 drop in each eye once daily at 9.00 pm (± 1 hour) for 3 months.
  Interventions: Drug: Lumigan 0.03% Unit Dose

INTERVENTIONS:
Drug: Monoprost — Monoprost®: Latanoprost 0.005% ophthalmic preparation is a sterile unpreserved oil-based solution for topical ophthalmic use. It is supplied in 0.30 ml single use polyethylene containers. The batch numbers and reanalysis dates will be stated in the certificate of analysis.
  Other Names: Latanoprost 0.005%
  Arms: Monoprost
Drug: Lumigan 0.01% — Lumigan® 0.01%: Bimatoprost eye drop solution is supplied in 3 ml multidose container.
  Other Names: Bimatoprost 0.1mg/ml
  Arms: Lumigan 0.01%
Drug: Lumigan 0.03% Unit Dose — Lumigan® 0.03% Unit Dose: Bimatoprost eye drop solution is supplied in 0.4 ml single use low density polyethylene (LDPE) containers.
  Other Names: Bimatoprost 0.3mg/ML
  Arms: Lumigan 0.03% Unit Dose

SUMMARY:
Primary objective:

The primary objective is to demonstrate the superiority of Monoprost® versus Lumigan® 0.01% and Lumigan® 0.03% Unit Dose in term of safety with respect to the assessment of conjunctival hyperaemia in the worse eye at Day 84.

The conjunctival hyperaemia will be scored using the MacMonnies photographic scale (0 to 5).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years old.
* Written informed consent.
* Association of the 3 following criteria:

  1. Both eyes have primary open angle glaucoma or ocular hypertension already treated and controlled by mono-therapy of Lumigan® 0.01% since at least 3 months (according to European Glaucoma Society guidelines).
  2. Intra Ocular Pressure ≤ 18 mm Hg in both eyes.
  3. With local intolerance signs in at least one eye defined by the association of:

3.1 Hyperaemia = Grade (2) or (3) or (4) following the photographic MacMonnies scale.

And 3.2.1 Presence of at least 2 symptoms with a level of severity ≥ 1 (= mild or moderate or severe) among the following 5 symptoms: irritation/burning, itching, tearing, eye dryness sensation, foreign body sensation.

And/Or 3.2.2 Presence of at least 2 signs with a level of severity ≥ 1 (= mild or moderate or severe) among the following 3 signs: superficial punctate keratitis, blepharitis, eyelid skin darkness.

Exclusion Criteria:

* - Presence of at least one severe objective sign among the following:

  * Global ocular staining with Oxford (0-15) grading scheme >12.
  * Blepharitis (Grade 4: Very severe, i.e. eczematiform lesion).
* Any ocular hypertension other than primary ocular hypertension or primary chronic open angle glaucoma (such as congenital, angle closure glaucoma, secondary glaucoma).
* Visual field not performed or not available within the 6 months before inclusion visit.
* Fundus not performed or not available within the 6 months before inclusion visit.
* Advanced stage of glaucoma:

  * Absolute defect in the ten degrees central point of the visual field.
  * Severe visual field loss according to the investigator's best judgement.
  * Risk of visual field worsening as a consequence of participation in the trial according to the investigator's best judgement.
* Best far corrected visual acuity ≤ 1/10.
* History of trauma, infection, inflammation within the 3 months before inclusion visit.
* Ongoing or known history of ocular allergy and/or uveitis and/or viral infection.
* Severe dry eye (defined by severe epithelial erosions of the cornea and/or use of dry eye medication with a frequency exceeding 8 instillations / day).
* Corneal ulceration.
* Palpebral abnormalities not related to medical treatment study and incompatible with a good evaluation.
* Any abnormality preventing accurate assessment e.g. reliable tonometry measurement, visual field examination.

Systemic/non ophthalmic/ exclusion criteria

* Non-controlled diabetic patient.
* Known or suspected hypersensitivity to one of the components of the study product.
* Any medical or surgical history, disorder or disease such as acute or chronic severe organic disease: hepatic, endocrine, neoplastic, haematological; immunosuppressive, infectious diseases, severe psychiatric illness, relevant cardiovascular abnormalities, etc… and/or any complicating factor or structural abnormality, judged by the investigator to be incompatible with the study.

Specific exclusion criteria for women

* Pregnancy, lactation.
* Childbearing potential woman who is not using a reliable method of contraception (oral contraceptive, intra-uterine device, subcutaneous contraceptive implant, vaginal ring, patch) and is not surgically sterilised.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Baudouin, Professor, Principal Investigator — Hopital des XV-XX
Locations (1):
- Laboratoires Théa, Clermont-Ferrand, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were enrolled at medical clinics from Dec 2013 to July 2016
Pre-assignment Details: the number of patients enrolled in 379 but as the primary Endpoint is Safety, the Baseline population is based on the safety Set and it corresponds to 373 patients
Groups:
- Lumigan 0.01% (Bimatoprost Eye Drop Solution): 1 drop in each eye once daily at 9.00 pm (± 1 hour) for 3 months.
  3-mL multidose containers
- Lumigan 0.03% UD (Bimatoprost Eye Drop Solution): one drop in each eye once daily at 9.00 pm (± 1 hour) in the inferior conjunctival cul-de-sac from D0 to D84.
  0.4-mL single-use low density polyethylene (LDPE) containers.
Period: Overall Study
Arm/Group | Monoprost | Lumigan 0.01% (Bimatoprost Eye Drop Solution) | Lumigan 0.03% UD (Bimatoprost Eye Drop Solution)
Started | 122 | 125 | 132
Completed | 106 | 113 | 117
Not Completed | 16 | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monoprost | Lumigan 0.01% | Lumigan 0.03% Unit Dose | Total
Number analyzed (Participants) | 119 | 124 | 130 | 373
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 44 | 48 | 138
  >=65 years | 73 | 80 | 82 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.9) | 67.4 (10.3) | 68.3 (10) | 67.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 78 | 218
  Male | 49 | 54 | 52 | 155
Region of Enrollment [Number; unit: participants]
  France | 24 | 25 | 26 | 75
  Germany | 14 | 12 | 15 | 41
  Spain | 50 | 52 | 51 | 153
  United Kingdom | 21 | 24 | 26 | 71
  Greece | 10 | 11 | 12 | 33

OUTCOME MEASURES:

1. Primary Outcome: Safety With Respect to the Assessment of Conjunctival Hyperaemia in the Worse Eye
Description: The primary endpoint is the change from baseline of conjunctival hyperaemia assessed on MacMonnies' 6 point ordinal scale, in the worse eye at the D84 visit. The primary statistical hypothesis tested is that Monoprost® is superior to Lumigan® 0.03% Unit Dose with regard to this primary endpoint, i.e. that in the worse eye the decrease from baseline in the MacMonnies 6 point ordinal scale is greater in the Monoprost® treated group than in the Lumigan® 0.03% Unit Dose group at the Day 84 visit.
  The conjunctival hyperaemia will be scored using the "McMonnies" photographic scale (0 to 5). The minimum score is 0 corresponding to a low hyperaemia and the maximum score is 5 corresponding to a higher hyperaemia.
  The Rows represent the number of participants with a change from Baseline to D84 corresponding to
  * "decrease of 3 points"
  * "decrease of 2 points"
  * "no change",
  * "increase of 2 points"
  * "increase of 1 point" on Mc Monnies scale
Time Frame: Day 84
Population: the primary analysis was performed in the mSAF.(All randomised patients of the Safety set with at least one eligible eye and with any safety information on treatment.)
Measure: Count of Participants; unit: Participants
Arm/Group | Monoprost | Lumigan 0.01% | Lumigan 0.03% Unit Dose
Number analyzed (Participants) | 112 | 118 | 124
Participants
  change at D84 -3 | 4 | 1 | 5
  change at D84 - 2 | 29 | 13 | 19
  change at D84 -1 | 47 | 59 | 42
  change at D84 0 | 29 | 39 | 38
  change at D84 +1 | 2 | 6 | 17
  change at D84 +2 | 0 | 0 | 1
  missing data | 1 | 0 | 2
Statistical Analysis 1: Comparison: Monoprost vs Lumigan 0.03% Unit Dose; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Monoprost vs Lumigan 0.01%; Test type: Superiority; p = 0.0045, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Monoprost | Lumigan 0.01% | Lumigan 0.03% Unit Dose
Serious Adverse Events (participants affected / at risk) | 3/119 | 2/124 | 2/130
Other Adverse Events (participants affected / at risk) | 0/119 | 0/124 | 0/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monoprost (N=119) | Lumigan 0.01% (N=124) | Lumigan 0.03% Unit Dose (N=130)
intervetebral disk protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
metastatic colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.